CLINICAL TRIAL: NCT04658901
Title: Endovenous Radiofrequency Closure Catheter and Endovenous Radiofrequency Closure Generator in the Treatment of Varicose Veins of Lower Extremity
Brief Title: ACOART RF CLOSURE:Radiofrequency for Varicose Veins of Lower Extremity in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acotec Scientific Co., Ltd (Industry)
Collaborators: Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACOART RF CLOSURE
Record Dates: First submitted 2020-11-04; First posted 2020-12-09 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-07

CONDITIONS: Varicose Veins of Lower Limb
Keywords: Varicose Veins of Lower Limb; radiofrequency ablation endovenous closure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): use endovenous radiofrequency closure catheter (ERA-C70,ERA-C30) and endovenous radiofrequency closure generator (ERA-G5) made by Acotec Scientific Co.,Ltd.
  Interventions: Device: ERA-C70,ERA-C30 and ERA-G5
- control group (Active Comparator): use the ClosureRFG™ and ClosureFast™ made by Medtronic Inc.
  Interventions: Device: ClosureFast™ and ClosureRFG™

INTERVENTIONS:
Device: ERA-C70,ERA-C30 and ERA-G5 — use endovenous radiofrequency closure catheter (ERA-C70,ERA-C30) and endovenous radiofrequency closure generator (ERA-G5) to treat varicose veins of lower extremity
  Arms: test group
Device: ClosureFast™ and ClosureRFG™ — use ClosureFast™ and ClosureRFG™ which has the indication of the treatment of varicose veins of lower extremity approved by NMPA
  Arms: control group

SUMMARY:
The purpose of the RCT trial is to determine whether endovenous radiofrequency closure catheter and endovenous radiofrequency closure generator is not inferior to ClosureFast™ and ClosureRFG™ in treating varicose veins of lower extremity.

DETAILED DESCRIPTION:
This trial is a prospective, multi-center, 1:1 randomized using endovenous radiofrequency closure catheter and endovenous radiofrequency closure generator versus ClosureFast™ and ClosureRFG™ to treat varicose veins of lower extremity. And parimary endpoint is Complete closure rate of great saphenous vein at 6 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years of age
* Patients clinically diagnosed as primary varicose great saphenous veins of lower extremity. And unilateral superficial varicose veins of lower extremity will be treated in this procedure.
* Patients with CEAP classification as C2-C5.
* Voluntarily participate in this study and sign the informed consent form

Exclusion Criteria:

* patients with target vein diameter < 2mm or > 15mm.
* the distance between the anterior wall of the vessel and the skin of the target vein under ultrasound is less than 0.5cm.
* patients with aneurysmal dilation at the saphenous femoral junction.
* patients with venous aneurysm (defined as venous hemangioma with a diameter greater than or equal to 2 times the diameter of the adjacent vein).
* thrombosis or thrombophlebitis in the trunk of great saphenous vein.
* the great saphenous vein is so tortuous that radiofrequency closure catheter cannot cross the vein trunk.
* patients with target diseased vessels who have received surgical treatment in the past.
* patients with deep venous thrombosis or a history of pulmonary embolism.
* patients with active implants such as pacemakers or ICD.
* patients with severe hepatic and renal dysfunction (ALT > normal upper limit 3 times; creatinine > 225umol/L).
* patients who are contraindications to anesthesia.
* patients with secondary varicose veins caused by deep venous thrombosis syndrome, Cockett syndrome (iliac vein compression syndrome), KT syndrome (venous malformation hypertrophy syndrome), arteriovenous fistula, etc.
* any serious or uncontrollable systemic disease (including uncontrolled hypertension, diabetes, active bleeding signs or severe coagulation disorders, etc.).
* patients with diseases that may cause difficulties in treatment and evaluation (such as malignant tumors, acute infectious diseases, septicemia, general intolerability of surgery, life expectancy less than 12 months, etc.).
* pregnant and lactating women, or those who had a planned birth during the study period.
* patients who have participated in clinical trials of other drugs or medical devices in the past 3 months.
* According to the judgement of the investigator, other situations that are not suitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-04-12 (Actual)

PRIMARY OUTCOMES:
Complete closure rate of great saphenous vein | at 6 months post-procedure
  Closure is defined as Doppler ultrasound examination (including color flow, compression, and pulsed Doppler) showing closure along the entire treated target vein segment with no discrete segments of patency exceeding 5 cm. Recanalization is defined as openings along the treated segment exceeding 5 cm in length as detected by duplex ultrasound.
  Complete closure rate = the number of subjects with closure of target vein in the group / the total number of subjects in the group x100%

SECONDARY OUTCOMES:
Device success rate | during procedure
  Device success is defined as the catheter could be advanced to the target position and retrieved successfully in the radiofrequency treatment procedure.
  Device success rate = the number of subjects with successful device in this group/the total number of subjects in this group x100%
Immediate technical success rate | during procedure (Instantly after the catheter retrieved)
  The technical success is defined as target vein closure. And closure is defined as Doppler ultrasound examination (including color flow,compression, and pulsed Doppler) showing closure along the entire treated target vein segment with no discrete segments of patency exceeding 5 cm. Recanalization is defined as openings along the treated segment exceeding 5 cm in length as detected by duplex ultrasound.
  Immediate technical success rate = the number of subjects successfully operated in this group/the total number of subjects in this group x100%
venous clinical severity score | at 6 months post-procedure
  Changes from baseline in venous clinical severity score (VCSS) (0-30, higher scores mean a worse outcome) in outpatient services. the VCSS was derived by the American Venous Forum from the CEAP classification and provides means by which clinical outcomes in venous disease can be monitored in time.Compared to the CEAP, VCSS is said to be more responsive to changes in disease severity, thus making it great for progressive rankings. It proved good inter and intra observer reproducibility and is often cited in quality of life assessments.
Aberdeen Varicose Vein Questionnaire | at 6 months post-procedure
  Changes from baseline in Aberdeen Varicose Vein Questionnaire (AVVQ) (0-33,higher scores mean a worse outcome) scores in outpatient services. The Aberdeen Varicose Vein questionnaire (AVVQ) with 14-question survey was used to determine the quality of life of patients with varicose veins both before and after surgery.
Evaluation of the use of devices | during procedure
  For endovenous radiofrequency closure catheter: evaluation on the degree of device flexibility, crossability, accuracy, usability (subjective evaluation scale: excellent, good and poor) For endovenous radiofrequency closure generator: evaluation on applicability,accuracy of identifying catheter version, stability in the procedure(subjective evaluation: yes or no)

CONTACTS AND LOCATIONS:
Overall Officials: Hongkun Zhang, MD, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital,Zhejiang University School of Medicine, Zhejiang, China